CLINICAL TRIAL: NCT06049823
Title: Comparison of Half- and Full-Grafting Alveolar Ridge Preservation With Different Sealing Materials: A Three-arm Randomized Clinical Trial
Brief Title: Alveolar Ridge Preservation With Different Grafting Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Choying Lin, assistent professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Chang Gung MH
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Bone Resorption
Keywords: alveolar ridge preservation; sealing material; resorbable membrane; non-resorbable membrane; dental implants
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The operator (L.C.Y.) was blinded to the assignment and opened the envelope just before the alveolar ridge preservation procedures, while both the participants and the examiners (C.M.Y., P.Y.K.) remained completely blinded to the assignments in the study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test1 (Experimental): half- (bottom 50% of socket filled with gelatin sponge and the top 50% of the socket filled with deproteinized bovine bone mineral mixed with collagen (DBBM-C)) then covered with a collagen membrane in tooth sockets
  Interventions: Procedure: Alveolar ridge preservation
- Test2 (Experimental): half- (bottom 50% of socket filled with gelatin sponge and the top 50% of the socket filled with deproteinized bovine bone mineral mixed with collagen (DBBM-C)) then covered with a nonresorbable membrane in tooth sockets
  Interventions: Procedure: Alveolar ridge preservation
- Control (Experimental): full-grafting (DBBM-C+ Collagen membrane) in tooth sockets
  Interventions: Procedure: Alveolar ridge preservation

INTERVENTIONS:
Procedure: Alveolar ridge preservation — Different grafting strategy of alveolar ridge preservation with different sealing materials

SUMMARY:
The aim of the present study was to compare the half-packed grafts that are covered with either a collagen or a nonresorbable membrane to the conventional alveolar ridge preservation procedures involving full-packed grafts and collagen membrane. The primary purpose was to evaluate the bone dimensional changes between the groups, and the secondary objective was to assess the potential contributing factors to clinical, radiographic and implant-related outcomes under different alveolar ridge preservation procedures.

DETAILED DESCRIPTION:
Regarding different surgical approaches in alveolar ridge preservation, limited studies directly compare collagen and non-resorbable membrane, and the comparison between half- and full- grafting strategy in clinical and radiographic outcomes was still lacking. The comparable effect of dimensional preservation between groups was shown except for more radiographic bone gain in full-grafting group. Contributing factors, including thin bone thickness , vertical root fracture related sockets, non-molar sites and large BPD might attenuate the effect of ARP. At implant placement, similar results in bone quality and keratinized mucosal width was found in all groups, while thicker vertical mucosal thickness was obtained when using nonresorbable membrane. All surgical modalities in alveolar ridge preservation yield stable peri-implant health 1 year after implant placement.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20 years old
2. presence of one or more hopeless teeth requiring extraction and subsequent implant placement due to reasons such as crack tooth, vertical root fracture, endodontic failure, unrestorable caries and severe periodontitis
3. the extraction socket should have more than two walls for ARP, which includes type I-II sockets (Palatal/ lingual defects were also included)
4. participants should have a stable periodontal condition or history of periodontitis that is well-controlled with good oral hygiene. The pocket depth of the adjacent tooth around the socket should be less than 3 mm as assessed with a periodontal probe (Hu-Friedy, Chicago, IL, USA).

Exclusion Criteria:

1. heavy smokers consuming more than half pack of cigarettes daily
2. women who were pregnant, lactating, or planning to be pregnant
3. history of psychiatric disorders
4. uncontrolled and complicated medical conditions that might hinder wound healing or bone metabolism, including poorly controlled diabetes, autoimmune disorders, receiving current radiotherapy in the head and neck regions, taking bisphosphonate and other antiresorptive agents.

Ages: 24 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
bone dimensional changes between the groups | 6-month healing period after alveolar ridge preservation
  Based on CBCT images, horizontal measurements by using AVIZO software (version 7.0, FEI). The measurements were repeated twice at a 2-week interval, and mean values were used for the final analysis (width or height in millimeters, mm):
  * Buccal bone plate thickness (BT) at 1 mm, 3mm, 5mm apical to the crest
  * Horizontal ridge width (HRW) at 1 at 1 mm, 3mm, 5mm apical to the crest
  * The change of HRW at 1, 3, 5 mm apical to crest (T2-T1).
  Vertical measurements in cross-sectional images:
  * Buccal bone height (BH)(mm)
  * Palatal/lingual bone height (PH)(mm)
  * The discrepancy between buccal and palatal/lingual height.(mm)
  * Midcrestal height (Mid-H)(mm)
  * The change of BH, PH, and Mid-H between immediate post-operative and 6 months later. (T2-T1)(mm).

SECONDARY OUTCOMES:
Clinical and implant related outcomes | 6-month healing period after alveolar ridge preservation
  Other clinical and implant-related parameters with descriptions:
  * Demographic data
  * Keratinized mucosal width (KMW)(mm)
  * Vertical mucosal thickness (VMT): measured from the mucosal profile to the crest of the ridge using a periodontal probe after buccal full-thickness flap elevation (Hu-Friedy, Chicago, IL, USA)(mm)
  * Bone density: Lekholm and Zarb's classification as types 1, 2, 3, or 4
  * Insertion torque: recorded once the implant was placed at the anticipated level with primary stability (NCM)
  * Marginal bone level change(mm) Based on the results of the normality tests, one-way ANOVA followed by the Tukey HSD or Kruskal-Wallis test with post hoc Dunn's test was performed for intergroup comparisons. The Chi-square association test (X2) was used to compare categorical variables between groups. Univariate linear regression methods were performed to investigate the factors to the changes of ridge width and height.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Chang Gung Memorial hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Raw data were generated at Taipei Chang Gung memorial hospital. Derived data supporting the findings of this study are available from the corresponding author(CYL) on request.

REFERENCES:
- [Derived] Hsieh CH, Kuo PY, Chiu MY, Lin CY. The Effectiveness of Different Grafting Strategies in Alveolar Ridge Preservation: A Retrospective Study of Two- and Three- Dimensional Radiographic Analysis. Int J Oral Maxillofac Implants. 2026 Jan 12;0(0):1-38. doi: 10.11607/jomi.11369. Online ahead of print. PMID 41525719
- [Derived] Lin CY, Chiu MY, Kuo PY, Wang HL. Half- and full-grafting alveolar ridge preservation with different sealing materials: A three-arm randomized clinical trial. Clin Implant Dent Relat Res. 2024 Jun;26(3):651-662. doi: 10.1111/cid.13327. Epub 2024 Apr 18. PMID 38638057